CLINICAL TRIAL: NCT04954417
Title: A Study on Vertebral Bone Strength by Micro-CT-Like Image: An Approach Based on Conditional Generative Adversarial Nets
Brief Title: A Study on Vertebral Bone Strength by Micro-CT-Like Image
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021179
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Deep Learning

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The vertebral specimens for this experiment were obtained from formalin-fixed human cadavers.The donors had dedicated their body for educational and research purposes to the local Institute of Anatomy prior to death, in compliance with local institutional and legislative requirements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MSCT image: Scanning of the vertebral body using MSCT
  Interventions: Diagnostic Test: Radiological scanning; Other: Deep learning; Procedure: Bio-mechanical testing
- micro-CT image: Scanning of the vertebral body using micro-CT
  Interventions: Diagnostic Test: Radiological scanning

INTERVENTIONS:
Diagnostic Test: Radiological scanning — The collected specimens subject to normalized Micro-CT and MSCT image acquisition, image reconstruction using standard algorithms, and bone structure observation using bone algorithms to obtain high-quality, standardized axial images.
Other: Deep learning — We will use a conditional generation adversarial network-based image mapping technique to train the mapping model between MSCT images and Micro-CT images, find the correspondence between the image information contained in each of MSCT and Micro-CT, and finally obtain high-resolution micro-CT-like images.
  Groups: MSCT image
Procedure: Bio-mechanical testing — we will cut a standardized cubic sample from the vertebral cancellous bone , obtain the bio-mechanical performance index of this cancellous bone sample by mechanical experiments, and analyze the correlation between bone structure of Micro-CT-like images and bio-mechanical index.
  Groups: MSCT image

SUMMARY:
In this study, we use conditional generation adversarial network to enhance the resolution of MSCT images and obtain micro-CT-like images. Based on this, we measure the bone structure indexes of micro-CT-like images and analyzed the correlation between bone structure and bio-mechanical indexes.

DETAILED DESCRIPTION:
In this study, we expect to collect 10 sets of vertebrae (between T6 and L5) from 10 formalin-fixed human cadavers. The study protocol was reviewed and approved by the local Institutional Review Boards.The collected specimens subject to normalized Micro-CT and MSCT image scanning, image reconstruction using standard algorithms, and bone structure observation using bone algorithms to obtain high-quality, standardized axial images. We will use a conditional generation adversarial network-based image mapping technique to train the mapping model between MSCT images and Micro-CT images, find the correspondence between the image information contained in each of MSCT and Micro-CT, and finally obtain high-resolution micro-CT-like images. After obtaining the Micro-CT-like images of the samples, we will segment and annotate the images (including different structures such as vertebral body, bone cortex) and train the Teacher-Student & U-Net++ deep learning architecture to achieve accurate segmentation of vertebral body regions, and obtain cancellous bone regions of interest. Based on this, we will analyze the bone structure characteristics of each spatial region in the images, including the thickness, spacing, orientation and distribution pattern of bone trabeculae and other indicators. Ultimately, we will cut a standardized cubic sample from the vertebral cancellous bone , obtain the bio-mechanical performance index of this cancellous bone sample by mechanical experiments, and analyze the correlation between bone structure of Micro-CT-like images and bio-mechanical index.

ELIGIBILITY:
Inclusion Criteria:

* We will collect human formalin-fixed vertebral specimens provided by the Department of Anatomy, Peking University School of Medicine. The expected number of enrolled specimens is approximately 100 vertebrae (between T6 and L5) .

Exclusion Criteria:

* The vertebrae with significant compression fractures, bone neoplasms, or other causes of significant bone destruction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The specimens for this experiment were obtained from formalin-fixed human cadavers.The donors had dedicated their body for educational and research purposes to the local Institute of Anatomy prior to death, in compliance with local institutional and legislative requirements.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Consistency or correlation | From the beginning of the experiment to 8 months
  Analyze the consistency or correlation between micro-CT and micro-CT-like bone structure indexes; analyze the correlation between micro-CT-like bone structure indexes and bio-mechanical indexes

CONTACTS AND LOCATIONS:
Overall Officials: huishu Yuan, Study Chair — Department of Radiology Peking University Third Hospital Beijing, China,
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No